CLINICAL TRIAL: NCT03733249
Title: Follow-up of Phase 1/2 Study of CaspaCIDe T Cells (BPX-501) From an HLA-partially Matched Family Donor After Negative Selection of TCR αβ+T Cells in Pediatric Patients Affected by Hematological Disorders
Brief Title: Long Term Follow-up Study for Patients Enrolled on the BP-004 Clinical Study
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-404
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Results first posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Acute Lymphoblastic Leukemia; Leukemia, Acute Myeloid (AML), Child; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Primary Immunodeficiency; Anemia, Aplastic; Hemoglobinopathies; Cytopenia; Fanconi Anemia; Diamond Blackfan Anemia; Thalassemia; Anemia, Sickle Cell
Keywords: Long term follow up; Gene-modified cells; ALL; AML; hematologic neoplasms; hematologic malignancies; anemia; congenital cytopenia; primary immune deficiencies; hemoglobinopathy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Primary Immunodeficiency Diseases; Anemia, Aplastic; Hemoglobinopathies; Cytopenia; Fanconi Anemia; Anemia, Diamond-Blackfan; Thalassemia; Anemia, Sickle Cell; Hematologic Neoplasms; Anemia | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rimiducid and Rivogenlecleucel (Experimental): Rimiducid: to treat uncontrolled GVHD in patients who have received rivogenlecleucel Rimiducid will be given at 0.4 mg/kg weight (intravenous infusion)
  No further rivogenlecleucel infusions are planned. Patients who received rivogenlecleucel in the BP-004 study will be evaluated for long-term safety and efficacy.
  Interventions: Drug: Rimiducid; Biological: rivogenlecleucel

INTERVENTIONS:
Drug: Rimiducid — Rimiducid is administered to treat chronic graft versus host disease
  Other Names: AP1903
Biological: rivogenlecleucel — donor T-cells modified with iCasp safety switch
  Other Names: BPX-501

SUMMARY:
This is a long-term follow up study evaluating the safety of BPX-501 T cells (rivogenlecleucel) and infused in pediatric patients previously enrolled on the BP-004 study.

DETAILED DESCRIPTION:
Subjects enrolled on the BP-004 study who have completed or discontinued from the study, and are beyond Day 180 will be requested to enroll on this long-term follow up protocol. Long term follow up for gene therapy clinical and safety endpoints will continue up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent by the patient or the patient's guardian for children who are minors
* Enrolled on BP-004 protocol, received BPX-501 infusion, completed or discontinued from the study, and are beyond Day +180.

Exclusion Criteria:

* Lack of parents'/guardian's informed consent for children who are minors
* Loss of allograft prior to 6 months

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 187 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals, Study Director — Bellicum Pharmaceuticals, Inc.
Locations (1):
- IRCCS Ospedale Pediatrico Bambino Gesù, Rome, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study BP-404 was the long-term follow-up for patients enrolled in the BP-004 study at the Italian site as well as patients in Saudi Arabia (patients enrolled and treated in the UK who moved back after hematopoietic stem cell transplantation. The below participant flow information pertains to all patients in the BP-004 study (NCT02065869)
Pre-assignment Details: 3 Enrolled patients did not undergo hematopoietic stem cell transplantation (HSCT)
Period: Overall Study
Arm/Group | Rimiducid and Rivogenlecleucel
Started (Patients receiving HSCT graft (HSCT Safety population)) | 184
Patients Receiving Rivogenlecleucel (BPX-501 Safety Population) | 171
Intent-to-Treat Population (Includes all patients treated with HSCT who received rivogenlecleucel at the dose of 1×10E6 cells/kg.) | 142
Patients Receiving at Least 1 Dose of Rimiducid | 16
Completed | 149
Not Completed | 35
Not completed — Death | 7
Not completed — Disease relapse | 16
Not completed — Lost to Follow-up | 4
Not completed — No rivogenlecleucel cells infused (non-evaluable) | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: HSCT safety population: All enrolled patients who received hematopoietic stem cell transplantation
Arm/Group | Rimiducid and Rivogenlecleucel
Number analyzed (Participants) | 184
Age, Continuous [Median (Full Range); unit: years] — Subject eligibility criteria: patients less than or equal to 18 years of age and greater than or equal to 1 month of age.
  years | 5.8 [0.1 to 18.1]
Age, Customized [Count of Participants; unit: Participants]
  < 2 years | 43
  2 to < 12 years | 105
  12 to ≤ 18 years | 35
  18 to ≤ 26 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 176
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 162
  More than one race | 1
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) in both malignant and non-malignant subpopulations at 1 and 2 years in the Intent-to-Treat (ITT) Population
Time Frame: 1 and 2 years after rivogenlecleucel infusion
Population: ITT Population: Includes all patients treated with HSCT who received rivogenlecleucel at the dose of 1×10E6 cells/kg
  Study BP-404 is the long-term follow-up study of patients of the BP-004 study who were enrolled at the Italian and Saudi Arabia sites. There is a second long-term follow-up study (BP-004 UK) for patients enrolled at the UK sites. The below results include data from both the BP-404 study and the BP-004 UK study. Individual results for either study are not available.
Measure: Count of Participants; unit: Participants
Groups:
- Malignant: Patients with malignant disease.
- Non-malignant: Patients with non-malignant disease.
Arm/Group | Malignant | Non-malignant
Number analyzed (Participants) | 62 | 80
Participants
  1 Year: Event Occurred | 8 | 3
  1 Year: Censored | 3 | 8
  1 Year: At Risk [Defined as: Total participants - (Event Occurred + Censored)] | 51 | 69
  2 Years: Event Occurred | 8 | 4
  2 Years: Censored | 4 | 13
  2 Years: At Risk [Defined as: Total participants - (Event Occurred + Censored)] | 50 | 63

2. Primary Outcome: Incidence of Disease-free Survival
Description: KM Parameter Estimates of disease-free survival (DFS) in the non-malignant subpopulation at 1 and 2 years in the Intent-to-Treat (ITT) Population
Time Frame: 1 and 2 years after rivogenlecleucel infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-malignant
Number analyzed (Participants) | 80
Participants
  1 Year: Event occurred | 4
  1 Year: Censored | 7
  1 Year: At Risk [defined as: Total participants - (Event occurred + Censored)] | 69
  2 Years: Event occurred | 5
  2 Years: Censored | 12
  2 Years: At Risk [defined as: Total participants - (Event occurred + Censored)] | 63

3. Primary Outcome: Relapse-free Survival
Description: Kaplan-Meier Parameter Estimates of Relapse-free survival rate (number of patients survived without experiencing a recurrence) at the 1-year and 2-year timepoints in the Intent-to-Treat (ITT) Population in the malignant study arm (patients with a malignant reason for their transplant).
  ITT Population: Includes all patients treated with HSCT who received rivogenlecleucel at the dose of 1×10E6 cells/kg
Time Frame: 1 and 2 years after rivogenlecleucel infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Malignant
Number analyzed (Participants) | 62
Participants
  1 Year: Event Occurred | 12
  1 Year: Censored | 0
  1 Year: At Risk | 50
  2 Years: Event Occurred | 13
  2 Years: Censored | 1
  2 Years: At Risk | 48

ADVERSE EVENTS:
Time Frame: BP-404 is the long-term follow-up study of patients in the BP-004 study who were enrolled at the Italian and Saudi Arabia sites. Since a summary of AEs is not available for the long-term studies alone, the below AE data pertain to Study BP-004 (AEs assessed up to180 days post rivogenlecleucel administration for serious AEs (including all-cause mortality) and 30 days post rivogenlecleucel for non-serious AEs [30 and 7 days post rimiducid administration for serious/non-serious AEs respectively]).
Groups:
- Rivogenlecleucel (BPX-501) Safety Population: All patients who received HSCT and went on to receive any dose of rivogenlecleucel.
- Rimiducid Safety Population: All patients who received at least 1 dose of rimiducid for the treatment of acute or chronic GvHD refractory to SoC treatment after rivogenlecleucel administration.
Arm/Group | Rivogenlecleucel (BPX-501) Safety Population | Rimiducid Safety Population
All-Cause Mortality (participants affected / at risk) | 7/171 | 0/16
Serious Adverse Events (participants affected / at risk) | 52/171 | 7/16
Other Adverse Events (participants affected / at risk) | 140/171 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivogenlecleucel (BPX-501) Safety Population (N=171) | Rimiducid Safety Population (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pneumopericardium (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Device damage (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 0
Acute graft versus host disease (Immune system disorders) | 4 | 2
Adenovirus infection (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 3 | 0
Device related infection (Infections and infestations) | 3 | 0
Encephalitis (Infections and infestations) | 2 | 0
Escherichia infection (Infections and infestations) | 2 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 2 | 0
Varicella zoster virus infection (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Juvenile chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Miller Fisher syndrome (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiopulmonary failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivogenlecleucel (BPX-501) Safety Population (N=171) | Rimiducid Safety Population (N=16)
Cytomegalovirus infection (Infections and infestations) | 34 | 0
Adenovirus infection (Infections and infestations) | 11 | 0
Human herpesvirus 6 infection (Infections and infestations) | 9 | 0
Acute graft versus host disease (Immune system disorders) | 48 | 3
Rash (Skin and subcutaneous tissue disorders) | 21 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 0
Diarrhea (Gastrointestinal disorders) | 20 | 0
Vomiting (Gastrointestinal disorders) | 20 | 0
Nausea (Gastrointestinal disorders) | 10 | 0
Pyrexia (General disorders) | 33 | 0
Chronic graft versus host disease (Immune system disorders) | 5 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Right ventricular failure (Cardiac disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT03733249/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT03733249/SAP_001.pdf